CLINICAL TRIAL: NCT05825989
Title: The Effects of Healthy Beat Acupunch on Physical Fitness of Thai Older Adults in Residential Homes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Siriluk Winitchayothin, RN, The Effects of Healthy Beat Acupunch on Physical Fitness of Thai Older Adults in Residential Homes, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB-NS2022/96.2811
Record Dates: First submitted 2023-03-14; First posted 2023-04-24 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Aging
Keywords: acupunch exercise; older adults; physical fitness; residential homes; cluster-randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Beat Acupunch Regimen (Experimental): The intervention group will receive the instructor-led HBA regimen 3 times/week for first 6 months, followed by the DVD-led HBA regimen for another 6 months.
  Interventions: Behavioral: Healthy Beat Acupunch Regimen
- Control group (No Intervention): The control group will continue their daily activities.

INTERVENTIONS:
Behavioral: Healthy Beat Acupunch Regimen — The Healthy Beat Acupunch (HBA) regimen, developed by Chen et al. (2017), is based on the Meridian Theory or Jing-Luo Theory. The HBA regimen focuses on body movement with hands swinging, resulting in the natural swinging of fists that hit on acupoints. There are three phases: phase 1 is activating qi and blood; phase 2 is punching meridians; phase 3 is relaxing body and mind.
  Other Names: Meridian cuffing
  Arms: Healthy Beat Acupunch Regimen

SUMMARY:
The purpose of this study is to test the effects of the first three months of instructor-led HBA regimen on physical fitness (aerobic endurance, lung capacity, upper body flexibility, lower body flexibility, handgrip strength, upper body strength, and lower body strength) between the HBA intervention and control groups, to test the effects of another three months of DVD-led HBA regimen followed by the three months of instructor-led on physical fitness between the HBA intervention and control groups and to test the changes at three and six months of the HBA regimen in comparison to the baseline of the physical fitness in the HBA intervention group.

DETAILED DESCRIPTION:
After the researcher meet the potential participants regarding the inclusion criteria, the researcher will inform purpose of study, human subjects protection, and termination in this study. Once participants receive all information and need to participate in this study, the researcher will ask permission participants to sign in their names in the informed consent and participant information sheet. If participants cannot sign their names, a thumbprint will be used instead of signatures. Therefore, the consent form will be completed by signatures or thumbprints.

This study will conduct in group exercise. The intervention group will receive the HBA program, 40 min/time, 3 times/week for 6 months. The control group will continue their routine activities of the residential homes.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate dependence or complete independence as defined by an Activity Daily Living assessment using the Barthel Index (BI Thai version) with a score of 61 or higher
* No cognitive impairment defined by a Short Portable Mental Status Questionnaire (SPMSQ Thai version) a score of ≥ 8
* No experience with the HBA regimen
* Able to communicate in Thai

Exclusion Criteria:

* Older adults whom physicians have advised not to exercise because of medical conditions, severe disease, such as severe cardiopulmonary disease (CVD, COPD), or severe musculoskeletal diseases, and have sensory impairments such as visual and auditory impairments.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical fitness: aerobic endurance | pretest (before receiving the HBA regimen)
  Aerobic endurance will be assessed by the 2 minutes step test. Participants will be asked to stand up in a straight position. The assessor marks the middle length between the patella and the pelvic bones at the wall with color tape. Participants raise their knees above the marked height as much as possible within 2 minutes. The score is the number of times the participants raise their knees above the marked height, which will be recorded.
Physical fitness: aerobic endurance | posttest 1 (after receiving the HBA regimen at 3 months)
  Aerobic endurance will be assessed by the 2 minutes step test. Participants will be asked to stand up in a straight position. The assessor marks the middle length between the patella and the pelvic bones at the wall with color tape. Participants raise their knees above the marked height as much as possible within 2 minutes. The score is the number of times the participants raise their knees above the marked height, which will be recorded.
Physical fitness: aerobic endurance | posttest 2 (after receiving the HBA regimen at 6 months)
  Aerobic endurance will be assessed by the 2 minutes step test. Participants will be asked to stand up in a straight position. The assessor marks the middle length between the patella and the pelvic bones at the wall with color tape. Participants raise their knees above the marked height as much as possible within 2 minutes. The score is the number of times the participants raise their knees above the marked height, which will be recorded.
Physical fitness: lung capacity | pretest (before receiving the HBA regimen)
  Lung capacity will be assessed by a TruZoneTM Peak Flow Meter. The TruZone will be reset to zero before participants hold the mouth-piece in their mouth. The score is the measurement of a deep breath, which is exhaled forcefully quickly in one out-breath. This will be recorded in liters.
Physical fitness: lung capacity | posttest 1 (after receiving the HBA regimen at 3 months)
  Lung capacity will be assessed by a TruZoneTM Peak Flow Meter. The TruZone will be reset to zero before participants hold the mouth-piece in their mouth. The score is the measurement of a deep breath, which is exhaled forcefully quickly in one out-breath. This will be recorded in liters.
Physical fitness: lung capacity | posttest 2 (after receiving the HBA regimen at 6 months)
  Lung capacity will be assessed by a TruZoneTM Peak Flow Meter. The TruZone will be reset to zero before participants hold the mouth-piece in their mouth. The score is the measurement of a deep breath, which is exhaled forcefully quickly in one out-breath. This will be recorded in liters.
Physical fitness: upper body flexibility | pretest (before receiving the HBA regimen)
  Upper body flexibility will be evaluated by a back scratch test. Participants raise their favored hand above the same shoulder and put their palm face down on their back with the fingers in a downward direction as much as possible. The other hand is placed palm up on the middle of the back as high as possible. The score is the distance in centimeters between the tips of the middle fingers, which will be recorded. If the tips of the middle fingers cannot touch, participants receive a minus score, if the middle fingers just touch a zero score is recorded, and if the tips of the middle fingers can overlap, participants receive a plus score.
Physical fitness: upper body flexibility | posttest 1 (after receiving the HBA regimen at 3 months)
  Upper body flexibility will be evaluated by a back scratch test. Participants raise their favored hand above the same shoulder and put their palm face down on their back with the fingers in a downward direction as much as possible. The other hand is placed palm up on the middle of the back as high as possible. The score is the distance in centimeters between the tips of the middle fingers, which will be recorded. If the tips of the middle fingers cannot touch, participants receive a minus score, if the middle fingers just touch a zero score is recorded, and if the tips of the middle fingers can overlap, participants receive a plus score.
Physical fitness: upper body flexibility | posttest 2 (after receiving the HBA regimen at 6 months)
  Upper body flexibility will be evaluated by a back scratch test. Participants raise their favored hand above the same shoulder and put their palm face down on their back with the fingers in a downward direction as much as possible. The other hand is placed palm up on the middle of the back as high as possible. The score is the distance in centimeters between the tips of the middle fingers, which will be recorded. If the tips of the middle fingers cannot touch, participants receive a minus score, if the middle fingers just touch a zero score is recorded, and if the tips of the middle fingers can overlap, participants receive a plus score.
Physical fitness: lower body flexibility | pretest (before receiving the HBA regimen)
  Lower body flexibility will be assessed by the chair sit-and-reach test. Participants sit on the front of a chair, then fully extend their right leg and place their foot up 90 degrees. Then, they move both hands to touch the big toe. The score is the distance in centimeters between the middle fingers of both hands and the big toe of the right foot, which will be recorded. Suppose their middle fingers cannot reach the big toe of the right foot. In that case, participants receive a minus score, if their middle fingers can reach the top of their big toe, a zero score is recorded, and if their middle fingers can reach or pass their big toe, participants receive a plus score.
Physical fitness: lower body flexibility | posttest 1 (after receiving the HBA regimen at 3 months)
  Lower body flexibility will be assessed by the chair sit-and-reach test. Participants sit on the front of a chair, then fully extend their right leg and place their foot up 90 degrees. Then, they move both hands to touch the big toe. The score is the distance in centimeters between the middle fingers of both hands and the big toe of the right foot, which will be recorded. Suppose their middle fingers cannot reach the big toe of the right foot. In that case, participants receive a minus score, if their middle fingers can reach the top of their big toe, a zero score is recorded, and if their middle fingers can reach or pass their big toe, participants receive a plus score.
Physical fitness: lower body flexibility | posttest 2 (after receiving the HBA regimen at 6 months)
  Lower body flexibility will be assessed by the chair sit-and-reach test. Participants sit on the front of a chair, then fully extend their right leg and place their foot up 90 degrees. Then, they move both hands to touch the big toe. The score is the distance in centimeters between the middle fingers of both hands and the big toe of the right foot, which will be recorded. Suppose their middle fingers cannot reach the big toe of the right foot. In that case, participants receive a minus score, if their middle fingers can reach the top of their big toe, a zero score is recorded, and if their middle fingers can reach or pass their big toe, participants receive a plus score.
Physical fitness: handgrip strength | pretest (before receiving the HBA regimen)
  Handgrip strength will be assessed by using a digital handgrip dynamometer. Participants hold the dynamometer with the fingers of their dominant hand and keep their arm parallel to the side of their body without moving the arm, then squeeze the holder for 3 seconds as hard as possible. Participants' handgrip strength will be measured two times. The score of the highest value will be recorded.
Physical fitness: handgrip strength | posttest 1 (after receiving the HBA regimen at 3 months)
  Handgrip strength will be assessed by using a digital handgrip dynamometer. Participants hold the dynamometer with the fingers of their dominant hand and keep their arm parallel to the side of their body without moving the arm, then squeeze the holder for 3 seconds as hard as possible. Participants' handgrip strength will be measured two times. The score of the highest value will be recorded.
Physical fitness: handgrip strength | posttest 2 (after receiving the HBA regimen at 6 months)
  Handgrip strength will be assessed by using a digital handgrip dynamometer. Participants hold the dynamometer with the fingers of their dominant hand and keep their arm parallel to the side of their body without moving the arm, then squeeze the holder for 3 seconds as hard as possible. Participants' handgrip strength will be measured two times. The score of the highest value will be recorded.
Physical fitness: upper body strength | pretest (before receiving the HBA regimen)
  Upper body strength will be assessed by a 60-second arm curl test. Participants sit on a chair and hold a dumbbell with their dominant hand (8-pound or 3.63 kilograms for men and 5-pound or 2.27 kilograms for women). Then, they lift the dumbbell up and down using the forearm repetitively. The score is the number of repetitions within 60 seconds, which will be recorded.
Physical fitness: upper body strength | posttest 1 (after receiving the HBA regimen at 3 months)
  Upper body strength will be assessed by a 60-second arm curl test. Participants sit on a chair and hold a dumbbell with their dominant hand (8-pound or 3.63 kilograms for men and 5-pound or 2.27 kilograms for women). Then, they lift the dumbbell up and down using the forearm repetitively. The score is the number of repetitions within 60 seconds, which will be recorded.
Physical fitness: upper body strength | posttest 2 (after receiving the HBA regimen at 6 months)
  Upper body strength will be assessed by a 60-second arm curl test. Participants sit on a chair and hold a dumbbell with their dominant hand (8-pound or 3.63 kilograms for men and 5-pound or 2.27 kilograms for women). Then, they lift the dumbbell up and down using the forearm repetitively. The score is the number of repetitions within 60 seconds, which will be recorded.
Physical fitness: lower body strength | pretest (before receiving the HBA regimen)
  Lower body strength will be assessed by the 60 seconds chair sit-to-stand test. Participants sit on the middle of the chair without an armrest or wheels. They put their feet on the floor equal width to their shoulder width. Then, they place both hands on their opposite shoulders. The score is the number of times that the subjects can stand up and sit down within 60 seconds, which will be recorded.
Physical fitness: lower body strength | posttest 1 (after receiving the HBA regimen at 3 months)
  Lower body strength will be assessed by the 60 seconds chair sit-to-stand test. Participants sit on the middle of the chair without an armrest or wheels. They put their feet on the floor equal width to their shoulder width. Then, they place both hands on their opposite shoulders. The score is the number of times that the subjects can stand up and sit down within 60 seconds, which will be recorded.
Physical fitness: lower body strength | posttest 2 (after receiving the HBA regimen at 6 months)
  Lower body strength will be assessed by the 60 seconds chair sit-to-stand test. Participants sit on the middle of the chair without an armrest or wheels. They put their feet on the floor equal width to their shoulder width. Then, they place both hands on their opposite shoulders. The score is the number of times that the subjects can stand up and sit down within 60 seconds, which will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Ban Bang Khae Social Welfare Development Center for Older Persons, Bang Khae, Bangkok
  - Watsanawet Social Welfare Development Center for Older Persons, Nakhon Luang, Phra Nakhon Si Ayutthaya

IPD SHARING:
Plan to Share IPD: No